CLINICAL TRIAL: NCT00914784
Title: The Incidence of Transfusion-Related Acute Lung Injury (TRALI) Following Blood Product Transfusion in Patients Undergoing Elective Orthopedic-Oncology Procedures
Brief Title: The Incidence of TRALI in Patients Undergoing Orthopedic-Oncology Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Idit Matot, Department of anesthesia and intensive care, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-IM-0295-CTIL
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Dyspnea; Pulmonary Edema
Keywords: TRALI; Transfusion; dyspnea; pulmonary infiltrates
MeSH Terms: conditions — Dyspnea; Pulmonary Edema; Transfusion-Related Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood from arterial line to test for PaO2
Oversight: Data Monitoring Committee: No

SUMMARY:
Currently Transfusion-related acute lung injury (TRALI) is the leading cause of transfusion-related mortality in the United States, and one of major post-transfusion complications. TRALI is defined as new ALI occurring within 6 hours from the onset of transfusion. It is manifested by acute dyspnea, hypoxemia and bilateral infiltrates in chest radiograph. TRALI may be caused by any blood product and is not dose-dependent. Associated risk factors include prolonged storage of blood products and underlying conditions such as severe IHD hematologic malignancies or active infections. Since TRALI has only recently been defined as a clinical entity, and its prevalence has been largely underestimated - the epidemiology of TRALI is not well established. Therefore the objective of this work is to study the incidence of TRALI in a patient population that receive blood products frequently, namely orthopedic-oncologic.

DETAILED DESCRIPTION:
Background

The transfusion of blood products is occasionally complicated by acute lung injury (ALI), which can progress to the acute respiratory distress syndrome (ARDS). Such transfusion-related acute lung injury, abbreviated TRALI, has been defined by both a National Heart, Lung, and Blood Institute (NHLBI) working group, and by a Canadian consensus conference (CCC), as new ALI occurring during or within six hours after a transfusion [1-2]. This definition is based entirely on clinical and radiological criteria and includes [2-4]:

1. ALI, as defined by [4]:

   A. The sudden onset of respiratory distress symptoms (dyspnea). B. Hypoxemia: as defined by a ratio of partial pressure of arterial oxygen to the fraction of inspired oxygen (PaO2/FiO2) below 300mmHg, or oxygen saturation (SpO2) below 90% on room air, or other clinical evidence of hypoxemia C. Bilateral infiltrates on frontal chest X-ray, without cardiomegaly. D. No clinical evidence of left atrial hypertension (congestive heart disease).
2. No preexisting ALI before transfusion.
3. During or within 6 hr after transfusion of any blood product.
4. No temporal relationship to an alternative risk factor for ALI. All types of blood products have been associated with TRALI, however, the plasma-rich components, such as fresh frozen plasma (FFP), whole blood, packed red blood cells (PC) and platelets, have been most frequently implicated [3, 5-10].

Prolonged storage of transfused products, use of FFP, and the presence of an underlying condition such as recent surgery, cytokine treatment, thrombocytopenia, massive blood transfusion, hematologic malignancies or cardiovascular disease requiring cardiopulmonary bypass (CABG) surgery, and active infection have been reported as risk factors for the development of TRALI [11-18].

The pathogenesis of TRALI involves the presence of anti-leukocyte antibodies and/or biologically active lipids from cell membrane fragments (and cytokines) in the donor's blood, triggering an inflammatory response within the recipient's pulmonary microvasculature, which in turn leads to lung injury [2,13,16,19-27].

The incidence of TRALI is not well established [28]. Nevertheless, using the NHLBI/CCC definition of TRALI, several retrospective studies reported the incidence of TRALI to be one case for every 1000-2400 units transfused [29-30]. This incidence estimate of 0.04% to 0.1% (or up to 0.85% among transfused patients) is comparable to other estimates from earlier studies that used older case definitions [6,12,31]. The only prospective cohort clinical surveillance study to use current diagnostic guidelines for TRALI reported an 8% incidence of TRALI in their intensive care unit (ICU) [32]. These data suggest that passive reporting systems greatly under-estimate the number of TRALI cases.

Even though underdiagnosed, TRALI is currently the leading cause of transfusion-related mortality in the United States [1,7,11]. The estimated mortality rate for recognized TRALI is 5%-8% [20]. However, most survivors recover completely with appropriate supportive care and can receive additional blood products in the future [11,20].

Due to the lacking epidemiology, and the increasing significance of TRALI as a major transfusion-associated complication, we stress the need for additional prospective surveillance studies.

Taken together, we wish to conduct a prospective observative study in order to evaluate the incidence of TRALI among patients undergoing elective orthopedic-oncology procedures. This patients' population receives blood product transfusions frequently, and may thus provide an adequate cohort for such study.

Study Objectives This work aims to study the prevalence of TRALI-associated morbidity and mortality in patients undergoing elective orthopedic-oncology procedures, and are transfused with blood products in the perioperative period.

In addition, we wish to evaluate whether:

A.The incidence of TRALI is higher in patients operated for malignancies (versus benign neoplasms) B.The incidence of TRALI is higher in patients treated with C.chemotherapy/radiation prior to surgery (versus non-treated) The incidence of TRALI is increasing with older blood products

Methods Study design An informed consent will be obtained from all orthopedic-oncology patients scheduled to have an elective surgery, except for those who require minor procedures (e.g., biopsies) which normally do not require transfusions. Diuretics and oral hypoglycemics will be discontinued the day prior to surgery, as dictated by the routines in our patients.

Peri-operative management Anesthetic and surgical management as well as blood product transfusion will adhere to standard practice.

Postoperatively, the patients will be transferred to the post-anaesthesia care unit and later to the orthopedic-oncology department, unless otherwise indicated.

In the postoperative period, departmental routines will guide blood product transfusions, pain management and fluid therapy.

Monitoring of patients who received transfusions

Every patient that receives blood products will be included in the study, whether it occurred pre-operatively, intra-operatively or post-operatively as long as they are hospitalized. For these patients we will document:

A.General demographics, including chronic diseases, medications and treatments (e.g., chemotherapy/radiotherapy).

B.Blood product information, including type, dosage and storage age. C.Intra- and post-operative data, including operative time, volume of crystalloids (and colloids) given during surgery and afterwards, urine output, the need for vasopressors, inotropes or diuretics, re-intubations, transfer to ICU and hospital length of stay (LOS).

For each unit of blood product transfused, we will commence patient monitoring for the next 6 hours. If several units are given in a sequel we will monitor the patient since the beginning of the first transfusion until 6 hours after the last transfusion. Monitoring will include:

1. Clinical symptoms of dyspnea.
2. PaO2/FiO2, or SpO2 on room air if arterial line is not obtainable - every 2 hours or when indicated by clinical signs.

   2.1. If PaO2/FiO2< 300mmHg, or SpO2< 90% on room air, or clinical signs of lung injury occur - chest X-ray will be obtained and diagnosed by two radiologists.
3. Hb (gr/dl) will be assessed according to the physician's decision.

Study size In the orthopedic-oncology department of Tel Aviv Sourasky Medical Center approximately 550 patients are operated annually, about 20% of whom receive transfusions. Accordingly, the study is planned for 5 years. Therefore the anticipated sample size is approximately 550 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years old, with ASA I-III, undergoing elective orthopedic-oncology procedures in the Sourasky Medical Center, and receiving blood products pre-, intra-, or post-operatively.

Exclusion Criteria:

* Patients with a history of chronic renal insufficiency (creatinine > 1.5 of normal value), congestive heart failure, hepatic dysfunction, preexisting ALI, or acute infection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged >18 years old, with ASA I-III, undergoing elective orthopedic-oncology procedures in the Sourasky Medical Center, and receiving blood products pre-, intra-, or post-operatively.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of TRALI in patients undergoing orthopedic-oncology procedures, following blood product transfusion | 2 years

SECONDARY OUTCOMES:
The correlation between the incidence of TRALI and the age of blood product | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, Study Chair — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel